CLINICAL TRIAL: NCT00972777
Title: A Study to Evaluate the Clinical and Microbial Efficacy of Besifloxacin Ophthalmic Suspension, 0.6% BID Compared to Vehicle in the Treatment of Bacterial Conjunctivitis.
Brief Title: Efficacy of Besifloxacin Ophthalmic Suspension in the Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 603
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-02

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besifloxacin (Experimental): 0.6% ophthalmic suspension
  Interventions: Drug: Besifloxacin
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle (Placebo)

INTERVENTIONS:
Drug: Besifloxacin — Besifloxacin 0.6% administered into the study eye two times a day for three days.
  Other Names: Besivance
  Arms: Besifloxacin
Drug: Vehicle (Placebo) — Vehicle administered to the study eye two times a day for three days.
  Arms: Vehicle

SUMMARY:
This study is being conducted to evaluate the clinical and microbial efficacy of besifloxacin ophthalmic suspension compared with vehicle in the treatment of bacterial conjunctivitis. This study was conducted as a phase IIb study and continued with further enrollment as a phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least one year of age.
* Subjects who have a clinical diagnosis of acute bacterial conjunctivitis.
* Subjects who are willing to discontinue contact lens wear for the duration of the study.

Exclusion Criteria:

* Subjects who have any uncontrolled systemic disease or debilitating disease.
* Subjects with known sensitivity or contraindications to besifloxacin, fluoroquinolones or any ingredients in study drugs.
* Subjects who are expected to require treatment with any disallowed medications.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Paterno, OD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

REFERENCES:
- [Derived] Haas W, Gearinger LS, Hesje CK, Sanfilippo CM, Morris TW. Microbiological etiology and susceptibility of bacterial conjunctivitis isolates from clinical trials with ophthalmic, twice-daily besifloxacin. Adv Ther. 2012 May;29(5):442-55. doi: 10.1007/s12325-012-0023-y. Epub 2012 May 25. PMID 22644963
- [Derived] DeLeon J, Silverstein BE, Allaire C, Gearinger LS, Bateman KM, Morris TW, Comstock TL. Besifloxacin ophthalmic suspension 0.6% administered twice daily for 3 days in the treatment of bacterial conjunctivitis in adults and children. Clin Drug Investig. 2012 May 1;32(5):303-17. doi: 10.2165/11632470-000000000-00000. PMID 22420526
- [Derived] Silverstein BE, Allaire C, Bateman KM, Gearinger LS, Morris TW, Comstock TL. Efficacy and tolerability of besifloxacin ophthalmic suspension 0.6% administered twice daily for 3 days in the treatment of bacterial conjunctivitis: a multicenter, randomized, double-masked, vehicle-controlled, parallel-group study in adults and children. Clin Ther. 2011 Jan;33(1):13-26. doi: 10.1016/j.clinthera.2010.12.004. PMID 21397770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two phase (IIB/III) integrated study. Phase IIb was conducted at 31 sites and Phase III at 28 sites in the United States. The first participant was enrolled in phase IIb on 10/30/2009, and last participant exited the study on 04/09/2010. Phase III enrolled its first participant on 04/05/2010 and last participant exited on 10/13/2010.
Pre-assignment Details: A total of 474 participants were enrolled in the integrated study in the intent to treat(ITT) population. 276 participants had culture confirmed bacterial conjunctivitis and were assigned to the modified intent to treat(mITT) population. 464 participants were assigned to the safety population. 446 participants completed the study.
Groups:
- Vehicle: Vehicle of besifloxacin ophthalmic suspension
Period: Overall Study
Arm/Group | Besifloxacin | Vehicle
Started | 231 | 243
Completed | 217 | 229
Not Completed | 14 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Physician Decision | 4 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Screening Failure | 2 | 1
Not completed — Missed visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besifloxacin | Vehicle | Total
Number analyzed (Participants) | 231 | 243 | 474
Age, Customized [Number; unit: participants]
  <2 years | 14 | 13 | 27
  2 - 11 years | 66 | 77 | 143
  12 - 17 years | 19 | 20 | 39
  18 - 29 years | 32 | 40 | 72
  30 - 39 years | 21 | 29 | 50
  40 - 49 years | 23 | 14 | 37
  50 - 59 years | 20 | 19 | 39
  >=60 years | 35 | 31 | 66
  Missing | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 133 | 275
  Male | 89 | 110 | 199
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 7 | 5 | 12
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 45 | 58 | 103
  White | 167 | 166 | 333
  Other | 4 | 5 | 9
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution
Description: The absence of both conjunctival discharge and bulbar conjunctival injection.
Time Frame: Visit 2
Population: Clinical Resolution at Visit 2, (LOCF), mITT Population.
Measure: Number; unit: eyes
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 135 | 141
eyes | 89 | 62

2. Primary Outcome: Microbial Eradication
Description: The absence of ocular bacteria that were present at or above pathogenic threshold levels at baseline.
Time Frame: Visit 2
Population: Microbial Eradication at Visit 2, (LOCF), mITT Population.
Measure: Number; unit: eyes
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 135 | 141
eyes | 115 | 77

3. Secondary Outcome: Clinical Resolution
Description: The absence of both conjunctival discharge and bulbar conjunctival injection.
Time Frame: Visit 3
Population: Clinical Resolution at Visit 3, (LOCF) mITT Population.
Measure: Number; unit: eyes
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 135 | 141
eyes | 103 | 94

4. Secondary Outcome: Microbial Eradication
Description: The absence of ocular bacteria that were present at or above pathogenic threshold levels at baseline.
Time Frame: Visit 3
Population: Microbial Eradication at Visit 3, (LOCF), mITT Population.
Measure: Number; unit: eyes
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 135 | 141
eyes | 115 | 91

ADVERSE EVENTS:
Time Frame: 7 days
Description: Safety Population, participants receiving at least one drop of study medication.
Arm/Group | Besifloxacin | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/228 | 0/236
Other Adverse Events (participants affected / at risk) | 0/228 | 0/236

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.